CLINICAL TRIAL: NCT06472284
Title: Train-of-four Monitoring Using the TetraGraph Neuromuscular Transmission Monitor to Evaluate Rocuronium Infusion Requirements During Major Neurosurgical and Surgical Procedures
Brief Title: TetraGraph in Rocuronium Infusions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00004154
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Rocuronium infusion (Experimental): Patients who are scheduled for elective, urgent or emergent surgery requiring the continuous infusion of the neuromuscular blocking agent, rocuronium.
  Interventions: Device: TetraGraph

INTERVENTIONS:
Device: TetraGraph — etraGraph is a unique, EMG-based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.

SUMMARY:
This is a prospective, non-blinded study to evaluate rocuronium infusion requirements using the TetraGraph Neuromuscular Transmission Monitor during surgical procedures in patients less than 18 yrs. of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years of age
* American Society of Anesthesiologists classification (ASA) 1-4
* Patients undergoing a surgical procedure with general anesthesia and requiring the continuous administration of rocuroniuim

Exclusion Criteria:

* Patients less than 28 days old
* Patients with history of a progressive or degenerative peripheral neurologic or neuropathic disorder
* Patients undergoing a surgical procedure in which neuromuscular blockade is not required
* Edematous patients

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
EMG changes | During the surgery (2-8 hrs.)
  Changes in the amplitude of the evoked response of the muscles
Maximum dose of rocuronium | During the surgery (2-8 hrs.)
  The maximum dose of rocuronium administered by a continuous infusion to maintain one twitch of the train of four (TOF)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided